CLINICAL TRIAL: NCT01053845
Title: Study of Integrity of Down Inhibitor Bundle at Patients Suffering of Neuropathic Pain
Acronym: PhyDoNe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0066; 2009-A00155-52 (Registry Identifier: ID RCB)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers; Patients Suffering of Peripheral Neuropathic Pain
Keywords: Neuropathic pain
MeSH Terms: conditions — Neuralgia

INTERVENTIONS:
Other: Neuropathic pain — to study the working of down inhibitor bundle at patients suffering of neuropathic pain

SUMMARY:
Several studies showed that activity of down inhibitor bundle is weakened in different painful pathologies as the fibromyalgy or the trigeminal nevralgy.

The purpose of the protocol is to study the working of down inhibitor bundle at patients suffering of neuropathic pain.

DETAILED DESCRIPTION:
Prospective study with comparison groups

ELIGIBILITY:
Inclusion Criteria:

* neuropathic patients group

  * Patient suffering of peripheral neuropathic pain
  * 18 years old women or men at least

Exclusion Criteria:

* • Healthy volunteers

  * 18 years old women or men at least

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the amplitude of N2P2 waves between healthy volunteers and patients suffering of peripheral neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France